CLINICAL TRIAL: NCT05872412
Title: Effect of Platinum-based Versus Non-platinum-based Neoadjuvant Chemotherapy in Triple-negative Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Mohammad Jahan Shams, Medical Officer, Department of Clinical Oncology, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BSMMU/2023/6669
Record Dates: First submitted 2023-05-14; First posted 2023-05-24 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Triple Negative Breast Cancer
Keywords: Triple negative breast cancer; Platinum; Neoadjuvant
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Doxorubicin; Cyclophosphamide; Paclitaxel; Carboplatin

STUDY DESIGN:
Intervention Model Description: This is a double-blinded randomized controlled trial to explore the efficacy and toxicity of platinum-based versus non-platinum-based neoadjuvant chemotherapy in triple-negative breast cancer.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platinum-based regimen (Experimental): Patients will be treated with doxorubicin 60 mg/m2 IV on day 1 and cyclophosphamide 600 mg/m2 IV on day 1 every 3 weeks for four cycles, followed by paclitaxel 80 mg/m2 IV weekly for 12 weeks concurrently with carboplatin (area under the curve: 6 mg/ml/min, i.v. every 3 weeks for four cycles).
  Interventions: Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Paclitaxel; Drug: Carboplatin
- Non-platinum based regimen (Active Comparator): Patients will be treated with doxorubicin 60 mg/m2 IV on day 1 and cyclophosphamide 600 mg/m2 IV on day 1 every 3 weeks for four cycles, followed by paclitaxel 80 mg/m2 IV weekly for 12 weeks.
  Interventions: Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Paclitaxel

INTERVENTIONS:
Drug: Doxorubicin — 60 mg/m2 IV bolus on day 1 every three weeks for four cycles.
  Other Names: Adriamycin
Drug: Cyclophosphamide — 600 mg/m2 IV over 1 hour on day 1 every three weeks for four cycles.
  Other Names: Cytoxan
Drug: Paclitaxel — 80 mg/m2 IV over 1 hour weekly for 12 weeks
  Other Names: Taxol
Drug: Carboplatin — Area under the curve: 6 mg/ml/min, i.v. every 3 weeks for four cycles
  Other Names: Paraplatin
  Arms: Platinum-based regimen

SUMMARY:
In this study, individuals with triple-negative breast cancer will receive either a platinum-based or non-platinum-based preoperative chemotherapy treatment. This study will help us identify which option is the most effective and safe.

DETAILED DESCRIPTION:
Breast cancer is a significant health concern, and triple-negative breast cancer (TNBC) is a particularly aggressive and lethal subtype. Chemotherapy is currently the only recommended systemic treatment for TNBC, with the standard regimen being a combination of anthracyclines and taxanes. Platinum agents have shown promising results in TNBC neoadjuvant chemotherapy due to their ability to damage DNA and be more effective in tumors with dysfunctional DNA repair mechanisms. However, there is still a lack of consensus on the optimal neoadjuvant chemotherapy regimen for TNBC. This study will be conducted to compare the responses and toxicities of platinum-based versus non-platinum-based neoadjuvant chemotherapy in TNBC patients receiving neoadjuvant chemotherapy in the Department of Clinical Oncology of Bangabandhu Sheikh Mujib Medical University (BSMMU), Shahbagh, Dhaka. After pretreatment evaluation, a total of 82 patients who fulfill the inclusion and exclusion criteria will be divided into Arm A and Arm B by simple random sampling. After the completion of the chemotherapy, all patients will undergo surgical management. A postoperative histopathology report will be collected and assessed by the investigator. During the treatment, the patients will be monitored before each cycle of chemotherapy, including physical examinations and laboratory investigations. All the relevant data will be compiled on a master chart first, and then statistical analysis of the results will be obtained by using Windows-based computer software facilities with Statistical Packages for Social Sciences. The data will be analyzed using the Chi-square test and the "T' test. The results will be presented in tables, figures, and diagrams. A significant value of 'p' will be decided at a level of 0.05 in two-tailed tests.

ELIGIBILITY:
Inclusion Criteria:

* Triple-negative breast cancer
* Stage II and III

Exclusion Criteria:

* Double primaries
* Male breast cancer
* Pregnant or lactating women
* Patients with Eastern Cooperative Oncology Group (ECOG) performance status more than two
* Patients below 18 years old
* Initial surgery of the primary site (excluding diagnostic biopsy)
* Serious concomitant medical illness including clinically significant cardiovascular disease
* Major surgery or trauma in the previous four weeks

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 82 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate | 1 year
  Pathological complete response: Post-operative pathology revealed no residual invasive cancer in the breast or lymph nodes.

SECONDARY OUTCOMES:
Clinical response | 1 year
  Clinical response will be assessed using the Response Evaluation Criteria in Solid Tumors (RECIST) criteria, which rely on a history, clinical exam, and imaging.
Treatment related acute toxicity | 1 year
  The American National Cancer Institute's "Common Terminology Criteria for Adverse Events" will be utilized to assess toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad J Shams, MBBS, MD, Principal Investigator — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] von Minckwitz G, Schneeweiss A, Loibl S, Salat C, Denkert C, Rezai M, Blohmer JU, Jackisch C, Paepke S, Gerber B, Zahm DM, Kummel S, Eidtmann H, Klare P, Huober J, Costa S, Tesch H, Hanusch C, Hilfrich J, Khandan F, Fasching PA, Sinn BV, Engels K, Mehta K, Nekljudova V, Untch M. Neoadjuvant carboplatin in patients with triple-negative and HER2-positive early breast cancer (GeparSixto; GBG 66): a randomised phase 2 trial. Lancet Oncol. 2014 Jun;15(7):747-56. doi: 10.1016/S1470-2045(14)70160-3. Epub 2014 Apr 30. PMID 24794243
- [Background] Zhang P, Yin Y, Mo H, Zhang B, Wang X, Li Q, Yuan P, Wang J, Zheng S, Cai R, Ma F, Fan Y, Xu B. Better pathologic complete response and relapse-free survival after carboplatin plus paclitaxel compared with epirubicin plus paclitaxel as neoadjuvant chemotherapy for locally advanced triple-negative breast cancer: a randomized phase 2 trial. Oncotarget. 2016 Sep 13;7(37):60647-60656. doi: 10.18632/oncotarget.10607. PMID 27447966
- [Background] Sikov WM, Berry DA, Perou CM, Singh B, Cirrincione CT, Tolaney SM, Kuzma CS, Pluard TJ, Somlo G, Port ER, Golshan M, Bellon JR, Collyar D, Hahn OM, Carey LA, Hudis CA, Winer EP. Impact of the addition of carboplatin and/or bevacizumab to neoadjuvant once-per-week paclitaxel followed by dose-dense doxorubicin and cyclophosphamide on pathologic complete response rates in stage II to III triple-negative breast cancer: CALGB 40603 (Alliance). J Clin Oncol. 2015 Jan 1;33(1):13-21. doi: 10.1200/JCO.2014.57.0572. Epub 2014 Aug 4. PMID 25092775
- [Background] Kumar P, Aggarwal R. An overview of triple-negative breast cancer. Arch Gynecol Obstet. 2016 Feb;293(2):247-69. doi: 10.1007/s00404-015-3859-y. Epub 2015 Sep 4. PMID 26341644
- [Background] Dent R, Trudeau M, Pritchard KI, Hanna WM, Kahn HK, Sawka CA, Lickley LA, Rawlinson E, Sun P, Narod SA. Triple-negative breast cancer: clinical features and patterns of recurrence. Clin Cancer Res. 2007 Aug 1;13(15 Pt 1):4429-34. doi: 10.1158/1078-0432.CCR-06-3045. PMID 17671126
- [Background] Jin J, Zhang W, Ji W, Yang F, Guan X. Predictive biomarkers for triple negative breast cancer treated with platinum-based chemotherapy. Cancer Biol Ther. 2017 Jun 3;18(6):369-378. doi: 10.1080/15384047.2017.1323582. Epub 2017 May 11. PMID 28494179
- [Background] Lips EH, Mulder L, Oonk A, van der Kolk LE, Hogervorst FB, Imholz AL, Wesseling J, Rodenhuis S, Nederlof PM. Triple-negative breast cancer: BRCAness and concordance of clinical features with BRCA1-mutation carriers. Br J Cancer. 2013 May 28;108(10):2172-7. doi: 10.1038/bjc.2013.144. Epub 2013 Apr 4. PMID 23558900
- [Background] Prat A, Cruz C, Hoadley KA, Diez O, Perou CM, Balmana J. Molecular features of the basal-like breast cancer subtype based on BRCA1 mutation status. Breast Cancer Res Treat. 2014 Aug;147(1):185-91. doi: 10.1007/s10549-014-3056-x. Epub 2014 Jul 22. PMID 25048467
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Telli ML, Hellyer J, Audeh W, Jensen KC, Bose S, Timms KM, Gutin A, Abkevich V, Peterson RN, Neff C, Hughes E, Sangale Z, Jones J, Hartman AR, Chang PJ, Vinayak S, Wenstrup R, Ford JM. Homologous recombination deficiency (HRD) status predicts response to standard neoadjuvant chemotherapy in patients with triple-negative or BRCA1/2 mutation-associated breast cancer. Breast Cancer Res Treat. 2018 Apr;168(3):625-630. doi: 10.1007/s10549-017-4624-7. Epub 2017 Dec 23. PMID 29275435